CLINICAL TRIAL: NCT06296030
Title: POOF: A Culturally Tailored Intervention for African American Trauma Based on Acceptance and Commitment Therapy
Brief Title: Culturally Tailored ACT for Black Trauma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Original PI, Dr. Jennifer Payne Shepard, transferred to another university. Study was discontinued.
Sponsor: Azusa Pacific University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0010
Record Dates: First submitted 2021-02-05; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Stress Disorders, Traumatic; Anxiety; Anxiety Disorders
MeSH Terms: conditions — Stress Disorders, Traumatic; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This project's research design is a two-by-two factorial design. Factor one, the type of ACT intervention delivered, has two levels - POOF delivery (level 1) and a classic ACT delivery (level 2). Factor two, the facilitator's first group treatment delivery, also has two levels. There are four (4) group facilitators. The first two facilitators deliver traditional ACT first (level 1), and the second two facilitators deliver POOF first (level 2). Each facilitator providing group treatment will facilitate two groups (classic and POOF), one after the next. However, facilitators will be randomized to the order in which they deliver their first group to reduce experimenter/ clinician history bias. All of the facilitators are licensed, mental health clinicians.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic ACT program (Experimental): Participants will engage in pre-test measures (anxiety, race-based stress, and psychological flexibility). Subjects will then participate in a 12-week telehealth group (once a week, 2 hours a week) with other group members where a classic Acceptance and Commitment Therapy protocol will be administered. After this, participants will engage in post-test measures.
  Interventions: Behavioral: Classic ACT program
- POOF ACT program (Experimental): Participants will engage in pre-test measures (anxiety, race-based stress, and psychological flexibility). Subjects will then participate in a 12-week telehealth group (once a week, 2 hours a week) with other group members where an Acceptance and Commitment Therapy protocol will be administered that has been culturally tailored to address African American racial trauma. After this, participants will engage in post-test measures.
  Interventions: Behavioral: POOF ACT program

INTERVENTIONS:
Behavioral: POOF ACT program — The goal of this study is to test this culturally tailored intervention (POOF) against classic ACT, to discover if POOF does better at decreasing race-based trauma in African Americans.Guided by the cultural humility framework and social determinants of health model, we examine POOF, a culturally-tailored ACT model for use with anxious African Americans. The POOF approach builds on research on ACT for the general population, an evidence-based intervention, by tailoring the language of ACT while retaining the fidelity of the ACT model. Our hypotheses examine acceptability and attitudes toward treatment, treatment outcomes for psychological symptoms (i.e., anxiety) and an ACT-related outcome (i.e., psychological flexibility), and a possible underlying mechanism of change (i.e., race-based stress).
  Other Names: POOF; Pulling Out Of Fire
  Arms: POOF ACT program
Behavioral: Classic ACT program — This protocol is for a classic, non-adapted ACT intervention.
  Other Names: Classic ACT; Traditional ACT
  Arms: Classic ACT program

SUMMARY:
Blacks in America more frequently meet the criteria for posttraumatic stress disorder (PTSD) than any other US race or ethnicity. Yet, blacks are among the groups least likely to use mental health services for trauma. Thus, a large number of traumatized blacks suffer silently and remain untreated.

Acceptance and Commitment Therapy (ACT) is an empirically-based psychological intervention that uses acceptance and mindfulness strategies, with commitment and behavior change strategies, to increase psychological flexibility and decrease anxiety outcomes. While culturally tailored mental health interventions have been shown useful for racial and ethnic minorities, there have been few efforts to tailor ACT for blacks. This NIH R21 would compare an ACT model specifically culturally tailored for blacks (POOF) to the classic ACT model in a randomized trial, where clinicians will conduct 12-session telehealth synchronous virtual groups. Eighty black participants who self-identify as suffering from stress or anxiety will be confidentially recruited. Two specific aims are proposed:

Aim 1) It is expected that POOF participants will report higher levels of acceptability of treatment than classic ACT participants and that POOF participants will have better adherence to treatment regimens than traditional ACT participants.

Aim 2) Given that race-based stress may mediate anxiety symptoms in U.S. based blacks, it is expected that POOF will decrease race-based stress, thereby mattering the most for improving anxiety outcomes for blacks.

The proposed R21 pilot study will be the first randomized controlled trial to evaluate an ACT intervention tailored explicitly for black racial trauma. This study will provide critical data needed to plan and design a future R01 controlled longitudinal effectiveness study. The long-term objective is to significantly reduce the prevalence of stress and anxiety-related symptoms due to traumatic events for Blacks by increasing treatment acceptability for this population. Since blacks have the highest rates of trauma prevalence and chronicity, yet they are still underrepresented in mental health treatment, this tailored intervention can have a significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* willing/ desiring to commit to engagement in a 12-week tele-health anxiety group
* self-identifies as African American or of Black American heritage
* age 18 years or over
* age 65 years or younger
* English-speaking, writing, and understanding
* able to provide informed consent
* is experiencing mild or moderate anxiety or stress-related symptoms, based on pre-screening testing
* has experience with video-based social media, Zoom, or other synchronous video-based modalities

Exclusion Criteria:

* At the screening, those who state they have additional psychological, behavioral, or medical disorders (outside of anxiety, stress, or trauma-related disorders) as their primary concern. For instance, if a participant was diagnosed with major depressive disorder as primary and an anxiety disorder as secondary, they would be excluded from the study.
* At the screening, those who are experiencing anxiety due to a physical condition (due to a cancer diagnosis or some other physical diagnosis) would be excluded from this study.
* Individuals who are experiencing extreme psychological symptoms are not appropriate for a tele-health group format.
* Persons who are on medication for any psychological disorder at the time of screening may not be appropriate for this tele-health group format.
* Those who have not been introduced to web-based formats of live interaction prior to the study (if they have no experience with technology or they are not comfortable with technology) would not be appropriate for this particular tele-health pilot study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Race-Based Traumatic Stress | 12-weeks
  The Race-Based Traumatic Stress Symptom Scale (RBTSSS)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Payne, Ph.D., Principal Investigator — Azusa Pacific University
Locations (1):
- Azusa Pacific University, Azusa, California, United States

IPD SHARING:
Plan to Share IPD: No